CLINICAL TRIAL: NCT07156825
Title: Methodological Guide for the Adaptation of Pediatric Speech Audiometry Tests Into Other Languages
Brief Title: Adaptation of Pediatric Speech Audiometry Tests Into Other Languages
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: Budapest University of Technology and Economics (Other)
Responsible Party: Principal Investigator, Dr. Gáborján Anita, M.D., Ph.D., Semmelweis University
Other Study IDs: SE 312/2021
Record Dates: First submitted 2025-08-06; First posted 2025-09-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss; Screening
Keywords: Audiometry, Speech; Speech Perception; Speech Reception Threshold Test; Speech Intelligibility; Speech; Auditory Threshold; Child, Preschool
MeSH Terms: conditions — Hearing Loss; Speech; Speech Intelligibility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1 N: Children 2 - 4,5 years of age; with normal hearing
- Group 2 N: Children 4,5 - 5,5 years of age; with normal hearing
- Group 3 N: Children 5,5 - 7 years of age; with normal hearing
- Group 1 P: Children 2 - 4,5 years of age; with impaired hearing
- Group 2 P: Children 4,5 - 5,5 years of age; with impaired hearing
- Group 3 P: Children 5,5 - 7 years of age; with impaired hearing

SUMMARY:
The objective of this study was to offer a comprehensive framework for the adaptation of speech audiometric tests into other languages. To date, this is the first universal protocol of its kind that systematically considers linguistic, phonological, and audiological aspects.

The present paper provides a protocol and an example for adaptation and standardization of the Mainzer Audiometric Test for Children (MATCH) to another language.

DETAILED DESCRIPTION:
To evaluate auditory function in children, speech audiometry is widely used in routine clinical settings across many countries. However, appropriate test materials are not available in several languages to date. Adapting a speech audiometry test to another language poses a significant challenge. The objective of this study was to offer a comprehensive framework for the adaptation of speech audiometric tests into other languages. To date, this is the first universal protocol of its kind that systematically considers linguistic, phonological, and audiological aspects.

The present paper is a methodological study for instrument translation; it provides a protocol and example for adaptation and standardization of the Mainzer Audiometric Test for Children (MATCH) to another language. The prospective adaptation process is divided into six phases: identifying test items and validating picture recognizability among children; ensuring linguistic conformity by comparing the phoneme distribution of the test vocabulary to spontaneous speech reference data; recording the speech material in a sound-treated environment following International Organization for Standardization (ISO) standards; equalizing the intelligibility of the recorded items through speech recognition testing in adults; standardizing the test on a cohort of normal-hearing children aged 3-6 years, stratified by age; finally, the diagnostic validity of the adapted test is evaluated by comparing speech recognition thresholds to pure-tone audiometry results in a clinical sample. Additionally, to determine sensitivity, specificity, and optimal cutoff points for detecting hearing loss, ROC analysis is used.

ELIGIBILITY:
Inclusion Criteria:

* Age: limits for age groups: 2-4,5; 4,5-5,5; 5,5-7, respectively.
* For control goups: normal hearing verified by pure tone audiometry and tympanometry
* For hearing-impairment groups: stable sensorineural hearing loss confirmed by audiological diagnostics

Exclusion Criteria:

* Children presenting with symptoms of upper respiratory tract infections
* Known speech-language developmental disorders
* Cognitive disorders

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 2-7, with normal hearing in case of control groups and with stable sensorineural hearing loss in case of hearing-impairment groups.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between SRTs obtained with the adapted MATCH and the PTA thresholds (500 Hz, 1, 2, and 4 kHz) | Through study completion, an average of 1 year.
  The primary outcome measure is the correlation between Speech Recognition thresholds obtained with the adapted MATCH and the Pure Tone Audiometry thresholds (500 Hz, 1, 2, and 4 kHz).

SECONDARY OUTCOMES:
Test-retest reliability (intraclass correlation coefficients, ICC) | Through study completion, an average of 1 year.
  Secondary outcome measures include test-retest reliability (intraclass correlation coefficients, ICC), to verify the reproducibility of the measurements.
Diagnostic performance | Through study completion, an average of 1 year.
  ROC analysis will be used to establish optimal cut-off points for clinical decision-making and to quantify the diagnostic performance of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Gaborjan, M.D., Ph.D., Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
It can be given out only in case of special request, with the permission of the study participants or their legal representatives.

REFERENCES:
- [Background] Schirkonyer V, Keilmann A, Harmuth C, Wachtlin B, Rader T, Bohnert A. The new Mainz speech test for children 3-7 years old (MATCH) : Design, standardization, and validation. HNO. 2020 Jan;68(Suppl 1):43-49. doi: 10.1007/s00106-019-00793-0. PMID 31915885

DOCUMENTS (3):
  • Study Protocol (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT07156825/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT07156825/SAP_001.pdf
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT07156825/ICF_002.pdf